CLINICAL TRIAL: NCT04740749
Title: Longevity, Functional Status and Quality of Life of the Compress® Compliant Pre-Stress System: a Prospective Study
Brief Title: Longevity, Functional Status and Quality of Life of the Compress® Compliant Pre-Stress System
Acronym: Compress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Masterthesis completed
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S64761
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-10

CONDITIONS: Compress Compliant Pre-Stress System; Malignant Bone Tumor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective group (Other): Patients who have to undergone the implant surgery
  Interventions: Device: Compress Compliant Pre-Stress System
- Retrospective group (Other): Patients that have already undergone the implant surgery
  Interventions: Device: Compress Compliant Pre-Stress System

INTERVENTIONS:
Device: Compress Compliant Pre-Stress System — Treatment of malignant femor tumors with the Compress Compliant Pre-Stress System

SUMMARY:
In the treatment of malignant bone tumors, it may be necessary to remove large areas of the femur. To replace these large parts of missing bone, a prosthesis can be used. One innovative technology developed by Biomet is the Compress® Compliant Pre-Stress System (CPS; Zimmer-Biomet, Warsaw, USA). This fixation device uses compression, via a short traction bar, to stimulate osteointegration at the bone-prosthetic interface, promote hypertrophy of the loaded bone, and avoid stress bypass of the host bone around a stiff intramedullary stem. Young patients cured of tumors have a long life expectancy and a compelling need for prosthetic fixation that is equally durable. Good bone fixation is a prerequisite for implant longevity.

Although the initial results are encouraging, there is a need for additional mid- to long-term survival data from larger patient series showing longevity of the system, as well as reporting of functional outcome. Furthermore, to the best of our knowledge, no study examining the survival of the device using prospective data already exists. In addition, no studies were found examining the quality of life of the patients with the CPS system.

DETAILED DESCRIPTION:
In the treatment of malignant bone tumors, it may be necessary to remove large areas of the femur. To replace these large parts of missing bone, a prosthesis can be used. One innovative technology developed by Biomet is the Compress® Compliant Pre-Stress System (CPS; Zimmer-Biomet, Warsaw, USA). This fixation device uses compression, via a short traction bar, to stimulate osteointegration at the bone-prosthetic interface, promote hypertrophy of the loaded bone, and avoid stress bypass of the host bone around a stiff intramedullary stem. Young patients cured of tumors have a long life expectancy and a compelling need for prosthetic fixation that is equally durable. Good bone fixation is a prerequisite for implant longevity. Since 1999, the CPS has been routinely placed on the orthopedics - UZ Leuven service and, as a result, more than 100 patients have been treated in this way. However, there are only few studies reporting on long-term performance of this system. In addition, limited data reporting functional outcome were found.

Although the initial results are encouraging, there is a need for additional mid- to long-term survival data from larger patient series showing longevity of the system, as well as reporting of functional outcome. Furthermore, to the best of our knowledge, no study examining the survival of the device using prospective data already exists. In addition, no studies were found examining the quality of life of the patients with the CPS system.

ELIGIBILITY:
Inclusion Criteria:

* Patients are/will be operated from 26/08/1999 onwards in UZ Leuven
* Implantation of the Compress Compliant Pre-Stress Device
* Informed consent obtained
* Patients are able to complete the questionnaires
* Age: minimum 7 years old

Exclusion Criteria:

* N/A

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Compress device survival | 25 years
  Revision will be used to determine implant survival. Revision will be defined as the explantation of any fixation mechanism: anchor plug, traction bar, spindle, sleeve, fixation pin

SECONDARY OUTCOMES:
Postoperative complications | 25 years
  Clinical assessment of postoperative complications. Complications will be classified acoording to Henderson classification.
Partial weight-bearing (crutches): duration | 25 years
  Clinical assessment to determine duration of partial weight-bearing
Radiography: signs of osseointegration | 25 years
  Radiographic assessment
EORTC Core Quality of Life questionnaire (QLQ-C30) | 25 years
  To assess the quality of life
Functional status | 25 years
  Musculoskeletal Tumor Society scoring system (MSTS) is used to determine the the physical and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Friedl Sinnaeve, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- KU Leuven/UZLeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No